CLINICAL TRIAL: NCT05017961
Title: Randomized Prospective Cohort Study Comparing Efficacy of Bone Marrow Aspirate Concentrate Combined With Cryopreserve Allograft Bone in the Treatment of Intra-Articular Calcaneal Fractures
Brief Title: Comparing Efficacy of Bone Marrow Aspirate Concentrate (BMAC) Combined With Allograft in Treatment of Calcaneus Fractures
Acronym: BMAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfortunately this study didn't receive funding.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Johnson, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003034
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Fractures, Bone
Keywords: calcaneus fracture; bone graft; bone marrow aspirate; stem cells
MeSH Terms: conditions — Fractures, Bone | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Autograft (Active Comparator): Following definitive fracture reduction a bone defect often remained in the substance of the calcaneus beneath the reduced posterior facet. In this group an autograft will be used to fill the void. For the purpose of autologous grafting, cancellous strips of bone will be harvested from the posterior superior iliac crest or proximal tibia. It shall be applied wherever bone loss exists as a result of the incident fracture or subsequent bone debridement(s). This will be the control arm.
  Interventions: Device: Autograft
- Allograft only (Other): Following definitive fracture reduction a bone defect often remained in the substance of the calcaneus beneath the reduced posterior facet. In this group a cryopreserved allograft bone (Musculoskeletal Tissue Foundation, New Jersey, NJ) will be used to fill the void. It shall be applied wherever bone loss exists as a result of the incident fracture or subsequent bone debridement(s).
  Interventions: Device: Allograft only
- Allograft combined with BMAC (Other): Following definitive fracture reduction a bone defect often remained in the substance of the calcaneus beneath the reduced posterior facet. In this group a cryopreserved allograft bone (Musculoskeletal Tissue Foundation, New Jersey, NJ) combined with BMAC will be used to fill the void. For the purpose of BMAC preparation, bone marrow will be collected from iliac crest or proximal tibia. It shall be applied wherever bone loss exists as a result of the incident fracture or subsequent bone debridement(s).
  Interventions: Device: Allograft combined with BMAC

INTERVENTIONS:
Device: Autograft — An autograft bone will be harvested from proximal tibia or posterior superior iliac crest. First the bony landmarks of the posterior iliac crest or proximal tibia are palpated. The skin is then injected down to and including the periosteum with 1% lidocaine without epinephrine. After 1 cm skin incision and gentle dissection of subcutaneous soft tissue, the bone harvesting device inserted through the skin and subcutaneous tissues until it reaches the cortical bone. Then, manual pressure is used to position the bone harvesting device against the dense cortical bone. A battery-powered power instrument is then will be used to drill the harvesting device into the medullary cavity. After the harvesting device insertion the cancellous strips of bone will be harvested and applied to the fracture site gap.At the conclusion of autograft bone harvesting procedure, the wound will be closed with 3-0 Nylon and a sterile dressing will be applied to the harvest site.
  Arms: Autograft
Device: Allograft only — The jar containing allograft tissue and cryopreservation solution will be placed in a sterile basin containing a warm (35°C to 39°C; 95°F to 102.2°F) sterile irrigant (Normal saline or 5% Dextrose in Lactated Ringer's Solution). The jar containing the allograft will remain in this solution until the contents of the jar flows freely upon inversion. The jar will be removed from the warm solution once free-flowing. Sterile gauze or the optional strainer will be used to decant the cryopreservation solution into a waste container. 5% Dextrose in Lactated Ringer's Solution will be added to the indicated fill line to immerse the allograft tissue. The cap will be replaced and inverted twice to suspend tissue until ready for use. 5% Dextrose will be decanted in Lactated Ringer's Solution prior to use. Implant will be used within 2 hours of thawing.
  Arms: Allograft only
Device: Allograft combined with BMAC — A bone marrow aspiration kit will be used for bone marrow aspiration. First the bony landmarks of the posterior iliac crest and sacroiliac joint are palpated. The skin is then injected down to and including the periosteum with 1% lidocaine without epinephrine. Then, the bone marrow aspiration trochar and needle are percutaneously inserted through the skin and subcutaneous tis- sues until it reaches the posterior iliac crest. The trajectory of the needle will be parallel to the iliac crest, or perpendicular to the Anterior Superior Iliac Spine (ASIS) or Posterior Superior Iliac Spine (PSIS), depending on the harvest site used. After the trochar is inserted into the posterior iliac crest but prior to aspiration, 1 mL of heparin (1,000 U/mL) will be preloaded into the syringe. Approximately 60 mL of bone marrow will be aspirated, which requires the use of two 30-mL syringes. At the conclusion of BMAC harvesting, a sterile dressing will be applied to the harvest site.
  Arms: Allograft combined with BMAC

SUMMARY:
The purpose of this study is to evaluate the efficacy of BMAC when used in conjunction with viable allograft bone for treating displaced intra-articular calcaneal fractures, in terms of rate of allograft incorporation into the host tissue, bone healing, and functional outcome.

DETAILED DESCRIPTION:
The study group will consist of patients with intra-articular calcaneal fractures admitted to our academic level I trauma center that underwent open reduction internal fixation. Inclusion criteria will be patients with a closed displaced intra-articular fracture Sanders type III without any evidence of neurovascular injury. Patients will be randomly divided into three groups according to the plan of management: autograft alone, viable allograft combined with BMAC, or viable allograft alone. Radiographic imaging and three-dimensional standing computed tomography will be used to assess the articular surface, Bohler's angle, the crucial angle of Gissane, and the height, width and length of the calcaneus. The American Orthopedic Foot and Ankle Society (AOFAS) ankle-hind-foot scoring system and visual analog scale (VAS) will be used to post-operative evaluation of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Closed displaced intra-articular fracture without any evidence of nerve or blood vessel injury, the fractures belonged to Sanders type III according to Sanders classification and amenable to open reduction internal fixation
* Life expectancy of at least 1 year
* Patient is willing to provide informed consent, is geographically stable and able to comply with the required follow up visits, testing schedule and medication regimen
* Adequate soft tissue coverage at the fracture site through primary closure.
* Unilateral or bilateral calcaneal fractures.

Exclusion Criteria:

* Pregnant or breastfeeding women or planning on becoming pregnant during the investigational period
* Patient is currently participating in an investigational drug or other device study or previously enrolled in this study.
* Uncontrolled diabetes mellitus (hemoglobin A1c levels > 10%)
* A current endocrine or metabolic disorder known to affect osteogenesis
* Currently has untreated malignant neoplasm(s), or is currently undergoing radiation therapy or chemotherapy.
* Inadequate neurovascular status in the involved limb that may jeopardize healing.
* Patients who have a preexisting calcaneus deformity that cannot accommodate a reduction or a previous history of osteomyelitis in the index limb.
* Other ipsilateral lower extremity fracture(s) if, in the opinion of the investigator, the treatment and/or rehabilitation of such fracture(s) will substantially interfere with the treatment, rehabilitation or other requirements outlined in this protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participant with satisfactory bone healing using American Orthopedics Foot and Ankle Society (AOFAS) ankle-hindfoot scoring system | baseline to 6 weeks
  The AOFAS ankle-hindfoot scoring system is the most commonly used instruments for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part. The scoring system range is from 0 to 100 with 100 being the best outcome score.
Percentage of participant with satisfactory bone healing using American Orthopedics Foot and Ankle Society (AOFAS) ankle-hindfoot scoring system | baseline to 12 weeks
  The AOFAS ankle-hindfoot scoring system is the most commonly used instruments for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part. The scoring system range is from 0 to 100 with 100 being the best outcome score.
Percentage of participant with satisfactory bone healing using American Orthopedics Foot and Ankle Society (AOFAS) ankle-hindfoot scoring system | baseline to 24 weeks
  The AOFAS ankle-hindfoot scoring system is the most commonly used instruments for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part. The scoring system range is from 0 to 100 with 100 being the best outcome score.
Percentage of participant with satisfactory bone healing using American Orthopedics Foot and Ankle Society (AOFAS) ankle-hindfoot scoring system | baseline to 52 weeks
  The AOFAS ankle-hindfoot scoring system is the most commonly used instruments for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part. The scoring system range is from 0 to 100 with 100 being the best outcome score.
Percentage of patient with satisfactory post treatment pain with Visual Analogue Scale (VAS) | baseline to 6 weeks
  The visual analogue scale or visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. Scale ranges from 0 to 10 with 10 being worse.
Percentage of patient with satisfactory post treatment pain with Visual Analogue Scale (VAS) | baseline to 12 weeks
  The visual analogue scale or visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. Scale ranges from 0 to 10 with 10 being worse.
Percentage of patient with satisfactory post treatment pain with Visual Analogue Scale (VAS) | baseline to 24 weeks
  The visual analogue scale or visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. Scale ranges from 0 to 10 with 10 being worse.
Percentage of patient with satisfactory post treatment pain with Visual Analogue Scale (VAS) | baseline to 52 weeks
  The visual analogue scale or visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. Scale ranges from 0 to 10 with 10 being worse.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Johnson, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No